CLINICAL TRIAL: NCT06911658
Title: Infectious Complications, Associated Factors, and Prognosis After Esophagectomy for Cancer: A French, Multicenter, Retrospective Study - CIFO-study
Brief Title: Infectious Complications After Esophagectomy
Acronym: CIFO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250038
Record Dates: First submitted 2025-03-13; First posted 2025-04-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Esophagectomy; Postoperative Complications; Infections; Pneumonia
Keywords: Postoperative infection; Esophagectomy complications
MeSH Terms: conditions — Postoperative Complications; Infections; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infectious complications represent the most common postoperative adverse events following esophagectomy for cancer, such as pneumonia (15% of cases). These complications increase immediate risks, lengthen hospital stays, and worsen patient quality of life.

The population includes patients admitted to intensive care after esophagectomy for cancer between January 1, 2017, and December 31, 2024.

The study focuses on this population due to the increasing incidence of esophageal cancer, the increased use of surgery for these indications, and the importance of postoperative infections in these complex procedures, despite their understudied nature in the current literature. Identifying modifiable risk factors could lead to corrective measures and thus improve the prognosis of postoperative patients.

The research focuses primarily on the incidence, types, factors, and prognosis associated with the occurrence of infections after esophagectomy for cancer. It also includes an analysis of the pathogens involved, their resistance profiles, and the antibiotic therapies used in first-line probabilistic treatment.

DETAILED DESCRIPTION:
The retrospective, multicenter study consists of the retrospective and pseudonymous collection of data from the medical reports of patients, covering the period from January 2017 to December 31, 2024, who were treated in each participating intensive care unit.

The investigators at each participating center will be responsible for screening and including patients, as well as obtaining their non-opposition.

Patients who were hospitalized for esophagectomy will be included, provided there are no exclusion criteria.

The following data will be collected after pseudonymization: only the first letter of the patient's last name and the first letter of their first name will be recorded, along with a study-specific coded number, which will differ for each center and indicate the order of inclusion of subjects. A correspondence table will be kept at each center for a period of 15 years. This table will be stored within each participating center.

At each participating center, data entry will be coordinated by the investigator responsible for the center. The collected data will be pseudonymized and stored in a secure database located at each participating center.

* If the patient is alive: the patient will be informed about the study. Data collection will begin only after the patient has been informed and only if the patient does not express opposition to the use of their data.
* If the patient is deceased and the vital status of the patient is known to the investigator: in this case, the investigator will verify in the patient's medical record that the patient has never expressed written opposition to the use of their data for research purposes. If the patient has never objected, their data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Underwent esophagectomy for cancer between January 1, 2017, and December 31, 2024
* Scheduled admission to intensive care for postoperative monitoring

Exclusion Criteria:

* Opposition to the use of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in intensive care unity.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of infections after esophagectomy for cancer | until the day 28

SECONDARY OUTCOMES:
Number of postoperative infectious episodes per participant, classified by anatomical site, as assessed retrospectively from hospitalization records | until the day 28
  Each infectious episode occurring within 28 days after esophagectomy will be retrospectively identified by review of hospitalization records. The anatomical site of infection (e.g., pulmonary, pleural, mediastinal, urinary, abdominal, surgical wound, bloodstream) will be determined based on the description found in medical documentation.
  The diagnosis of infection will rely on retrospective analysis of recorded clinical signs (e.g., fever), laboratory data (e.g., leukocytosis, elevated CRP), imaging reports (e.g., CT scan, chest X-ray), and physician assessmentsdocumented in the medical file.
  The unit of measure is : number of infectious episodes per participant. The data will be reported as the total number of episodes and their distribution by anatomical site, summarized per participant and overall using descriptive statistics (median [IQR], counts, percentages).
Presence of predefined pathogens during postoperative infectious episodes, as assessed retrospectively from hospitalization records | until the day 28
  For each postoperative infectious episode occurring within 28 days after esophagectomy, the presence or absence of specific pathogens will be retrospectively extracted from hospitalization reports using a structured checklist.
  The pathogens are not recorded as free-text entries but as binary variables (Yes/No) based on the presence of documentation in medical reports (microbiology results, discharge summaries, etc.).
  The predefined list includes :
  * Gram-positive cocci : Streptococcus spp., Enterococcus spp., E. faecium, Staphylococcus aureus (including MRSA)
  * Gram-negative bacteria : Haemophilus spp., Enterobacteriaceae (groups 1-3), non-fermenting bacilli (P. aeruginosa, A. baumannii, S. maltophilia)
  * Resistance profiles : ESBL-producing Enterobacteriaceae, carbapenemase-producing organisms
  * Fungi : Yeasts
  * Polymicrobial vs. monomicrobial infections Only pathogens explicitly mentioned in the clinical documentation (culture or PCR results) are recorded. The data are collected usi
Association between preoperative and perioperative clinical variables and the occurrence of postoperative infection, as assessed by multivariable logistic regression analysis of hospitalization records | until the day 28
  This outcome aims to explore the association between clinical and surgical factors and the risk of developing at least one infectious episode within 28 days following esophagectomy.
  Postoperative infections will be identified retrospectively based on hospitalization records. A multivariable logistic regression analysis will be conducted, with infection occurrence (Yes/No) as the dependent variable.
  Covariates will include :
  * Demographic characteristics : age and sex
  * Lifestyle factors : tobacco use and alcohol consumption (>2 drinks/day)
  * Nutritional status and general severity : Body Mass Index (BMI), IGS2 score at ICU admission
  * Comorbidities : cardiovascular disease (hypertension, myocardial infarction, congestive heart failure), chronic pulmonary disease, cerebrovascular disease (including stroke or transient ischemic attack), peripheral vascular disease (including aortic aneurysm >6 cm), diabetes (complicated or not), renal failure, liver disease (moderate or severe), dementi
Occurrence of major complications (sepsis, septic shock, AKI, ARDS, or death) within 28 days after esophagectomy, as documented in hospitalization records, compared between infected and non-infected patients | until day 28
  Association between postoperative infection and the occurrence of major complications (sepsis, septic shock, AKI, ARDS, or death), as assessed by logistic regression analyses of hospitalization records.
  Description
  This outcome assesses the relationship between the occurrence of postoperative infection (within 28 days of esophagectomy) and the development of the following complications :
  * Sepsis (according to Sepsis-3)
  * Septic shock (according to Sepsis-3)
  * Acute kidney injury (AKI according to KDIGO)
  * Acute respiratory distress syndrome (ARDS according to the Berlin's definition)
  * Mortality All events will be collected retrospectively from hospitalization records. A logistic regression will be used for each outcome separately to estimate the effect of infection (Yes/No) on the likelihood of each complication.
  Unit of measure : Odds Ratio (OR) with 95% Confidence Interval for each complication
Association between postoperative infection and length of hospital stay, as assessed by linear regression analysis of hospitalization records | until day 28
  Length of hospital stay (in days, from surgery to discharge) will be extracted from hospitalization records.
  A linear regression model will be used to assess whether the occurrence of a postoperative infection is associated with a prolonged hospital stay, adjusted for relevant covariates.
  Unit of measure : Median difference in number of days, with 95% Confidence Interval

CONTACTS AND LOCATIONS:
Overall Officials: François DEPRET, MD-PHD, Principal Investigator — APHP; DEPRET, Principal Investigator — APHP
Locations (2):
- France (2):
  - Hôpital Saint-Louis - APHP, Paris
  - Saint Louis Hospital, Paris

IPD SHARING:
Plan to Share IPD: No